CLINICAL TRIAL: NCT04207177
Title: Immunosuppressive Drugs and Gut Microbiome: Pharmacokinetic- and Microbiome Diversity Effects
Acronym: MicrobioTac
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Anders Åsberg, Head of Laboratory, Oslo University Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MicrobioTac-MPA
Record Dates: First submitted 2019-12-17; First posted 2019-12-20 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Kidney Transplant; Complications; Immune Suppression
MeSH Terms: interventions — Mycophenolic Acid; Tacrolimus

STUDY DESIGN:
Intervention Model Description: The main study is based on treatment allocation outside of thsi protocol but a subgroup of living donor recipients will be randomized to wither one week tacrolimus or mycophenolate mofetil treatment before transplantation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mycophenolate mofetil (Active Comparator): In the subgroup of living donor recipients included before transplantation this group will be treated with mycophenolate mofetil (750 mg BID) for one week
  Interventions: Drug: Mycophenolate Mofetil 500 mg Tab
- Tacrolimus (Active Comparator): In the subgroup of living donor recipients included before transplantation this group will be treated with tacrolimus (BID, dose by weight) for one week
  Interventions: Drug: Tacrolimus capsule

INTERVENTIONS:
Drug: Mycophenolate Mofetil 500 mg Tab — Twice daily dosing of MMF only for a week before transplantation in this subgroup. All patients will get maintenance treatment With MMF in combination With tacrolimus and steroids after transplantation.
  Other Names: MMF-arm
  Arms: Mycophenolate mofetil
Drug: Tacrolimus capsule — Twice daily dosing of tacrolimus only for a week before transplantation in this subgroup. All patients will get maintenance treatment With tacrolimus in combination With MMF and steroids after transplantation.
  Other Names: Tac-arm
  Arms: Tacrolimus

SUMMARY:
Kidney transplant recipients of living- and deceased donor grafts and treated with both mycophenolate mofetil (MMF) and tacrolimus (Tac) will be included. A 12-hour pharmacokinetic (PK) investigation of both mycophenolate (MPA) and Tac will be performed in pharmacokinetic steady state conditions between 3 to 8 weeks and one year after transplantation. Feces samples will be collected before (if possible), 1 week after transplantation and at the day of the 12-hour PK investigations. Data on dietary intake and physical activity will be obtained in association with the feces sampling in all patients. Patients will be invited to a follow-up visit one year after transplantation where the 12-hour PK investigation, feces sampling, dietary and activity data collection is repeated. Standard follow-up data after renal transplantations, such as acute rejection episodes, infections, renal function, post transplant diabetes mellitus (PTDM), protocol biopsies, adherence to immunosuppressive drugs, graft loss and death will be collected for all patients up to 5 years after transplantation according to standard schedule at the transplant center.

A subgroup of kidney transplant recipients scheduled for living donor transplantation will be included before transplantation for pre-transplant investigations in addition to the investigations after transplantation. These patients will be randomized to either receive one week of treatment with MMF or Tac before transplantation. Feces samples and a 12-hour PK investigation will be performed after one week of treatment (before transplantation).

DETAILED DESCRIPTION:
The analyses of feces samples will be performed by utilizing shotgun, next generation sequencing in order to determine the bacterial, fungal sand viral microbiome. Drug concentrations will be analyzed with high performance Liquid chromatography With double mass spectrometry detector (HPLC-MS/MS) technology and both free and total plasma MPA concentrations, total mycophenolate glucoronide (MPAG) concentrations and total whole blood Tac and methylated Tac-metabolite concentrations will be determined.

ELIGIBILITY:
Inclusion Criteria:

* De novo standard risk kidney transplant recipients.
* Patients scheduled to receive tacrolimus and mycophenolate mofetil as part of their immunosuppressive therapy following transplantation (clinical decision not influenced by this study).
* First kidney transplant only.
* Adult patients.

Exclusion Criteria:

- Pregnant or lactating female patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-10-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
investigate the association between microbiome diversity and 12-hour mycophenolate area under the curve (AUC) | 1 year
  Association between microbiome diversity measures and AUC of mycophenolate for a dose interval (AUC0-tau)
investigate the association between microbiome diversity and 12-hour mycophenolate Maximum concentration (Cmax) | 1 year
  Association between microbiome diversity measures and Cmax of mycophenolate

SECONDARY OUTCOMES:
association between microbiome diversity and 12-hour tacrolimus AUC | 1 year
  Association between microbiome diversity measures and AUC0-tau of tacrolimus
effects of mycophenolate mofetil treatment on gut microbiome changes in treatment naïve patients and associated mycophenolate AUC changes | 1 week
  Changes in microbiome diversity measures and mycophenolate AUC0-tau, with one week of mycophenolate mofetil treatment.
investigate the effects of tacrolimus treatment on gut microbiome changes in treatment naïve patients and associated tacrolimus AUC changes | 1 week
  Changes in microbiome diversity measures and tacrolimus AUC0-tau with one week of tacrolimus treatment
investigate if Torque Teno Virus (TTV) is a clinical useful "immunometer", i.e. reflect overall immunosuppression of the recipient | 1 year
  Associations between TTV viral load (DNAemia) and acute rejection episodes (biopsy proven)
Association between microbiome diversity measures and Cmax of tacrolimus | 1 year
  Association between microbiome diversity measures and Cmax of tacrolimus
Association between microbiome diversity measures and absolute bioavailability (F) of tacrolimus | 1 year
  Association between microbiome diversity measures and F of tacrolimus
effects of mycophenolate mofetil treatment on gut microbiome changes in treatment naïve patients and associated mycophenolate Cmax changes | 1week
  Changes in microbiome diversity measures and mycophenolate Cmax with one week of mycophenolate mofetil treatment.
effects of mycophenolate mofetil treatment on gut microbiome changes in treatment naïve patients and associated mycophenolate time to Cmax (Tmax) changes | 1week
  Changes in microbiome diversity measures and mycophenolate Tmax with one week of mycophenolate mofetil treatment.
effects of mycophenolate mofetil treatment on gut microbiome changes in treatment naïve patients and associated mycophenolate time to terminal phase elimination rate constant (kel)changes | 1 week
  Changes in microbiome diversity measures and mycophenolate kel with one week of mycophenolate mofetil treatment.
effects of tacrolimus treatment on gut microbiome changes in treatment naïve patients and associated tacrolimus time to Cmax (Tmax) changes | 1 week
  Changes in microbiome diversity measures and tacrolimus Cmax with one week of tacrolimus treatment.
effects of tacrolimus treatment on gut microbiome changes in treatment naïve patients and associated tacrolimus time to Cmax (Tmax) changes | 1 week
  Changes in microbiome diversity measures and tacrolimus Tmax with one week of tacrolimus treatment.
effects of tacrolimus treatment on gut microbiome changes in treatment naïve patients and associated tacrolimus time to terminal phase elimination rate constant (kel) changes | 1 week
  Changes in microbiome diversity measures and tacrolimus kel with one week of tacrolimus treatment.
investigate if Torque Teno Virus (TTV) is a clinical useful "immunometer", i.e. reflect overall immunosuppression of the recipient | 1 year
  Associations between TTV viral load (DNAemia) and opportunistic vial infections in need of drug treatment
investigate if Torque Teno Virus (TTV) is a clinical useful "immunometer", i.e. reflect overall immunosuppression of the recipient | 1 year
  Associations between TTV viral load (DNAemia) and opportunistic bacterial infections requiring hospitalization

OTHER OUTCOMES:
integrate the updated knowledge on mycophenolate and tacrolimus pharmacokinetics following renal transplantation in a combined population pharmacokinetic model for individualized dosing | 1 year
  Relative predictive error (PE%) of the developed pharmacokinetic model
integrate the updated knowledge on mycophenolate and tacrolimus pharmacokinetics following renal transplantation in a combined population pharmacokinetic model for individualized dosing | 1 year
  Relative root mean squared error (RMSE%) of the developed pharmacokinetic model

CONTACTS AND LOCATIONS:
Overall Officials: Karsten Midtvedt, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
Not allowed by Norwegian Law to share data without specific contract. Upon contact With the responsible investigator it is however possible to share data under a specified contract